CLINICAL TRIAL: NCT04593420
Title: Treatment of Aggressive Prostate Cancer in Real Life: Initiation, Schedule and Management of Triptorelin Treatment.
Acronym: TALISMAN
Status: Completed | Type: Observational
Sponsor: Ipsen (Industry)
Responsible Party: Sponsor
Other Study IDs: A-FR-52014-241
Record Dates: First submitted 2020-10-13; First posted 2020-10-20 (Actual); Last update posted 2022-12-21 (Actual); Status verified 2022-12

CONDITIONS: Prostate Cancer
MeSH Terms: conditions — Prostatic Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

SUMMARY:
The purpose of the protocol is to describe the proportion of subjects treated continuously with triptorelin during 12 months following treatment initiation. This study will take place at 187 locations (approximately) in France.

ELIGIBILITY:
Inclusion Criteria:

* At least 18 years old
* Histologically confirmed prostate cancer
* Triptorelin to be initiated in its labelled indication for a planned total duration of at least 12 months; decision to start triptorelin was made voluntarily by the physician as part of routine medical practice, prior to the inclusion in the study
* Ability to understand and complete questionnaire,

Exclusion Criteria:

* Previously received a hormonal therapy during the last 6 months before inclusion,
* Simultaneously participates in a clinical trial.

Min Age: 18 Years | Sex: Male
Age Groups: Adult, Older Adult
Study Population: 786 subjects presenting a prostate cancer histologically confirmed and eligible to start triptorelin treatment for at least 12 months will be included in the study. They should also be able to complete a self-questionnaire.
Sampling Method: Probability Sample
Enrollment: 817 (Actual)
Dates: Start 2020-11-30 (Actual); Primary Completion 2022-12-08 (Actual); Study Completion 2022-12-08 (Actual)

PRIMARY OUTCOMES:
Proportion of subjects treated continuously with triptorelin for the 12 months | 12 months
  The proportion of subjects treated continuously with triptorelin for the 12 months following treatment initiation, with any formulation and any route of administration. The treatment status (i.e. patient continuously treated / patient not continuously treated) will be assessed according to the investigator's judgment.

SECONDARY OUTCOMES:
Planned total duration of triptorelin treatment | Baseline, 6 months, 12 months
Primary reasons of choice of planned total triptorelin treatment duration | baseline, 6 month, 12 months
  Description of the primary reason of choice of planned total triptorelin treatment duration declared by the investigator, at V1; and at V2 and V3 if the planned total duration is modified.
Parameters that influence the planned total duration of triptorelin treatment | Baseline
  Identification of parameters that influence the planned total duration of triptorelin treatment including but not limited to the following parameters: Circumstance of prescription, Prostate Cancer (PCa) aggressiveness criteria, Prior PCa treatments, Concomitant PCa treatments, Subject's characteristics: age, weight, Karnofsky score, specific comorbidities and concomitant treatments, genetic predisposition.
Parameters that influence the modification of the planned total duration of triptorelin treatment | 12 months
  Identification of parameters that influence the modification (if any) of the planned total duration of triptorelin treatment including but not limited to the following parameters: PCa aggressiveness criteria at 12 months (PSA, concomitant treatments for prostate cancer, symptoms, metastases assessment), Subject's characteristics: age, weight, Karnofsky score, specific comorbidities and concomitant treatments, genetic predisposition at baseline, follow up assessments, care pathway.
Formulation and administration route of triptorelin prescribed | baseline, 6 and 12 months
  Formulation and administration route of triptorelin prescribed (monthly intramuscular, 3-monthly subcutaneous, 3-monthly intramuscular, 6-monthly intramuscular).
Description of the reasons of choice of formulation and administration route of triptorelin prescribed | baseline
  monthly intramuscular, 3-monthly subcutaneous, 3-monthly intramuscular, 6-monthly intramuscular) at V1, according to the investigator.
Parameters that influence the choice of formulation and administration route of triptorelin prescribed | baseline
  Identification of parameters that influence the choice of formulation and administration route of triptorelin prescribed (monthly intramuscular, 3-monthly subcutaneous, 3-monthly intramuscular, 6-monthly intramuscular) at V1 including but not limited to the following parameters: Disease with symptoms, total planned duration of treatment, highly evolutive disease, heavy PCa concomitant treatment, physical frailty of subjects, psychological context of subjects, potential impact on compliance, subject afraid of injection, anticoagulant treatment, BMI, Preferred investigator formulation/route
Description and change at each follow-up visit from baseline | baseline, 6 months, 12 months
  Description and change at each follow-up visit (V2, V3) from baseline (V1) in each of the 6 sub-scales of the QLQ-PR25 questionnaire (urinary symptoms, incontinence aid, bowel symptoms; treatment related symptoms, sexual activity, sexual functioning). QLQ-PR25 score is distributed from 1 (not at all) to 4 (very much).

CONTACTS AND LOCATIONS:
Overall Officials: Ipsen Medical Director, Study Director — Ipsen
Locations (1):
- Ipsen Central Contact, Paris, France

IPD SHARING:
Plan to Share IPD: Yes
Qualified researchers may request access to patient level data and related study documents including the clinical study report, study protocol with any amendments, annotated case report form, statistical analysis plan, and dataset specifications. Patient level data will be anonymized and study documents will be redacted to protect the privacy of study participants.
  Any requests should be submitted to www.vivli.org for assessment by an independent scientific review board.
Time Frame: Where applicable, data from eligible studies are available 6 months after the studied medicine and indication have been approved in the US and EU or after the primary manuscript describing the results has been accepted for publication, whichever is later.
Access Criteria: Further details on Ipsen's sharing criteria, eligible studies and process for sharing are available here (https://vivli.org/members/ourmembers/).
URL: https://vivli.org/members/ourmembers/

REFERENCES:
- [Derived] Lebret T, Crehange G, Pello-Leprince-Ringuet N, Perrot V, Rigaud J. Treatment of aggressive prostate cancer with triptorelin in real life in France: the TALISMAN study. Ther Adv Urol. 2025 Oct 15;17:17562872251382970. doi: 10.1177/17562872251382970. eCollection 2025 Jan-Dec. PMID 41122488